CLINICAL TRIAL: NCT01131247
Title: PHASE II CLINICAL PROTOCOL FOR THE TREATMENT OF PATIENTS WITH RELAPSED/REFRACTORY CHRONIC LYMPHOCYTIC LEUKEMIA WITH A COMBINATION OF BENDAMUSTINE AND OFATUMUMAB
Brief Title: PH2 Trial in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL) With a Combination of Bendamustine & Ofatumumab
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Nevada Cancer Institute (Other)
Collaborators: Cephalon (Industry); GlaxoSmithKline (Industry)
Responsible Party: Mark Kirschbaum, MD, Nevada Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVCI 09-15; 18083/6265 (Other: Cephalon)
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: CLL; bendamustine; ofatumumab; blood cancer; leukemia; lymphoma; lymphocyte; refractory; Advanced; relapsed; hematologic; hematology; antibody; non-Hodgkin lymphoma; small lymphocytic lymphoma; nevada cancer institute; cephalon; Glaxosmithkline
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Neoplasms; Leukemia; Lymphoma; Recurrence; Lymphoma, Non-Hodgkin | interventions — ofatumumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ofatumumab + bendamustine (Experimental)
  Interventions: Drug: ofatumumab + bendamustine

INTERVENTIONS:
Drug: ofatumumab + bendamustine — Loading dose of ofatumumab at 300mg IV with subsequent doses at 100mg IV on D1 of all cycles (maximum of 6 cycles) in combination with bendamustine 90mg/m2 on day 2 of all cycles. Neulasta 6mg SQ will also be given on day 8 of cycle 1 only.
  Other Names: Ofatumumab / Brand: Arzerra; Bendamustine / Brand: Treanda

SUMMARY:
Investigational Drugs:

Ofatumumab (Azerra) + bendamustine (Trenda)

Route of Administration:

Intravenous (IV)

Hypothesis:

This study is designed to assess the toxicity and overall response rate. Ofatumumab is a fully human monoclonal antibody (A type of protein made in the laboratory that can bind to substances in the body, including tumor cells) that shows promising activity in the treatment of CLL as a single agent. It is thought that by combining it with Bendamustine, an FDA approved treatment for CLL, the effect on CLL will be greater than if Ofatumumab is given alone. Ofatumumab is FDA approved for the treatment of relapsed/refractory CLL.

Participation:

Approximately 37 relapsed/refractory CLL subjects will participate in this study over two years.

Treatment Plan:

A maximum of 6 cycles of treatment will be allowed. During day 1 of cycle 1 ofatumumab IV 300mg will be administered. On day 1 of all cycles ofatumumab treatment will be followed by bendamustine IV 90mg/m2. On day 2 of all cycles, bendamustine IV 90mg/m2 will be administered. On day 3 of all cycles, neulasta SQ 6mg will be given. On day 8 of cycle 1 only patients will receive ofatumumab IV 1000mg. During cycles 2 through 6 ofatumumab 1000mg will be given on day 1 only.

Follow-up:

Patients will be followed monthly for six months, then every three months for five years then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Must be >/= 18 years old and able to provide consent
* Must have diagnosis of CLL as defined by NCI criteria
* Must require chemotherapy
* Must be previously treated with a minimum of one course of prior chemo or other treatment
* Serum creatinine <1.8 mg/dl
* Bilirubin must be </= 2 mg/d, unless secondary to tumor
* Must have adequate liver function (as defined as <2x ULN, unless related to CLL)
* AST/ALT <2x ULN
* Performance status 0-2
* Women of child bearing age must be willing to use accepted/effective method of birth control.

Exclusion Criteria:

* Not have received prior treatment with cytotoxic chemotherapy or immunotherapy.
* Not have autoimmune hemolytic anemia or autoimmune thrombocytopenia
* Not have history of corticosteroid treatment for CLL
* Not have CNS disease
* Not have clinically significant infections
* Patients with a second malignancy, other than basal cell carcinoma of the skin or in situ carcinoma of the cervix are not eligible.
* Not have positive serology for Hepatitis B or Hepatitis C
* Not have be known to be HIV positive
* Not have New York Classification III or IV hear disease

Other protocol specific criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate/ Efficacy
  The primary objective for this trial is to evaluate the overall response rate (CR+PR) of bendamustine and ofatumumab in patients with relapsed/refractory CLL.

SECONDARY OUTCOMES:
Safety Evaluation
  The first secondary objective is to evaluate the toxicity of patients with relapsed/refractory CLL treated with bendamustine and ofatumumab.
Response Rate
  Other secondary objectives include: evaluating the complete response rate, progression-free survivial, overal survival and time to next therapy
Correlative Analysis
  This study also aims to determine whether expression of of ZAP-70, CD38, IgVH status, and chromosomes, correlate with response rate, duration of response, and survival

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kirschbaum, MD, Principal Investigator — Nevada Cancer Institute; Jose Leis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, PHoenix/Scottsdale, Arizona, United States

REFERENCES:
- See also: Visit Nevada Cancer Institute Website for more information on investigator or trial — http://www.nevadacancerinstitute.org/